CLINICAL TRIAL: NCT00152568
Title: The Effectiveness of Car Seat Checks at Routine Pediatric Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11119A
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Car Seat Check

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Child Passenger Safety Technician services (Experimental)
  Interventions: Behavioral: Car Seat Check (behavior)

INTERVENTIONS:
Behavioral: Car Seat Check (behavior) — At time of well child visit, family receives the services of a certified child passenger safety technician, including assessment, car seat distribution if needed and training.

SUMMARY:
The purpose of this research is to evaluate the effectiveness of checking car seats during pediatric well-child visits on the use and properness of use of car seats for children 0-8 years. We are following up with families when they return for the next pediatric check up to see if they are appropriately using car seats for their children.

DETAILED DESCRIPTION:
The purpose of this investigation is to evaluate the effectiveness of a car seat inspection at the time of a pediatric visit on the proper use of car seats 4-6 months later.

Motor vehicle-related injury is the leading cause of death of children. Proper restraint in a motor vehicle reduces the risk of fatality in a crash by approximately 70%. However, multiple studies have found approximately 85% of car seats are misused. Urban poor and minority populations have been found to have higher child passenger death rates, and may have lower car seat usage rates than the rest of the population. Child passenger safety (CPS) technicians trained by the National Highway Traffic Safety Administration (NHTSA) and certified by the American Automobile Association (AAA) capably check proper car seat usage in "check up" events, and operate recently established "fitting stations." However, we are not aware of an attempt to provide the CPS technical services to families attending a routine checkup with their medical provider.

This project will involve implementing and evaluating a program providing car seat checks at the time of routine pediatric visits at the Friend Family Health Center (FFHC). To determine if the car seat checks improve proper car seat use, children who receive the intervention will have their car seat use reassessed at the time of a scheduled return visit to their medical provider. The frequency of routinely scheduled health maintenance visits is greatest for the youngest children. Opportunities to collect follow up car seat use data therefore will be greatest for the youngest children. This evaluation will focus on 0 year olds. While we will also assess the older children and booster seat use, the sample size calculation for this study was determined for these younger children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-8 years
* Child's family has a vehicle

Exclusion Criteria:

* Children over 8 years of age
* Child's family does not have a vehicle

Max Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 364 (Actual)
Dates: Start 2001-06; Primary Completion 2003-09 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Car seat us | median of 105.5 days

SECONDARY OUTCOMES:
Proper car seat use | 86.5 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyran Quinlan, M.D., M.P.H., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Grossman DC, Garcia CC. Effectiveness of health promotion programs to increase motor vehicle occupant restraint use among young children. Am J Prev Med. 1999 Jan;16(1 Suppl):12-22. doi: 10.1016/s0749-3797(98)00120-2. PMID 9921382